CLINICAL TRIAL: NCT01921244
Title: Shared Decision Making to Improve Care and Outcomes for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: FP00005038
Record Dates: First submitted 2013-08-05; First posted 2013-08-13 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Autistic Disorder; Pervasive Developmental Disorder; Child Development Disorders, Pervasive; Asperger Syndrome; Autism Spectrum Disorder; Autism
Keywords: Autistic Disorder; Decision Making; Medication Therapy Management
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive; Asperger Syndrome; Autism Spectrum Disorder | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Approximately 120 families will be asked to participate as "usual care" subjects and will complete surveys before and immediately after their visit, and approximately 3 months after the visit. These families will not receive the decision aid nor will their provider have been trained how to use the decision aid. All participating providers will have up to 10 "usual care" patients enrolled at baseline prior to allocation. During the trial, the control group ["usual care" providers] will have up to 10 additional patients enrolled for ongoing "usual care" data collection. After the trial is complete, the control group providers will cross over to the intervention arm.
- Intervention (Experimental): Approximately 80 families/patients with regularly scheduled clinic follow-up visits in the Division of Developmental and Behavioral Pediatrics (DDBP) at Cincinnati Childrens with providers trained on shared decision making will receive the decision aid prior to their index visit and complete surveys before and immediately after their visit, and approximately 3 months later.
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — Parents will receive an intervention modified from the previously published tool called "Autism: Should My Child Take Medicine for Challenging Behavior?" This packet provides parents with educational information, elicits parent ratings of particular behavioral domains, describes behaviors that are and are not amenable to medication treatment, and elicits parent preferences regarding treatment. Providers will be trained on use of the intervention in practice to promote shared decision making during clinical encounters.
  Other Names: Use of Medication to Treat Challenging Behavior in Autism
  Arms: Intervention

SUMMARY:
Children with Autism Spectrum Disorder (ASD) commonly experience behavioral challenges that may be improved with pharmacotherapy, including difficulties with sleep, attention, hyperactivity, impulsivity, anxiety, obsessive-compulsive behavior, mood swings, self-injury, and aggression. While 34-58% of children with ASD take medication for such behaviors, there is wide practice variation nationally and a lack of evidence to support the use of most commonly prescribed agents. Complex clinical situations such as this where there is no clear "best choice" regarding which behaviors to target and which medications to use lend themselves well to the use of a Shared Decision Making (SDM) tool to ensure that well-informed parent preferences shape every treatment plan.

The primary goal of this study is to modify a previously published decision aid about use of medication to manage challenging behaviors in children with autism to make it easy to implement in practice and then evaluate this version in terms of proximal decisional outcomes and parent/child outcomes 3 months later. Providers in a Developmental-Behavioral Pediatric clinic will be enrolled and randomly allocated to intervention or control (treatment as usual) groups. Initially, providers randomized to the intervention group will test and refine the modified intervention. Once the intervention is finalized, eligible patients of participating providers will be enrolled in the randomized controlled trial to test the efficacy of the intervention. Following the trial, control group providers will be crossed over and receive the intervention. Both proximal decisional outcomes (e.g. parent decisional conflict, provider amount of SDM, parent knowledge of treatment options) and outcomes 3 months later (e.g. parenting stress, decisional conflict, and change in child behavioral symptoms) will be assessed.

Approximately 10 providers and 240 of their patients with autism will be included in the study. Chart reviews, parental surveys, and recordings of provider-parent-patient interactions during the index visit will be collected at baseline (prior to physician allocation), during the intervention trial, and after the control group has crossed over. Between- and within-group analyses will examine factors associated with parental decisional conflict and whether the intervention produces significant improvements in outcomes over and above typical autism care. Analyses will include multiple linear regression modeling and general linear models / repeated measure models, accounting for data clustered by provider.

DETAILED DESCRIPTION:
SDM involves clinicians sharing information about treatment options and parents sharing their goals, concerns, and preferences to ensure that treatment plans are based on what matters most to well-informed parents. SDM often incorporates use of decision aids, which are balanced sources of information about treatment options for a particular condition. Decision aids consistently increase knowledge, improve treatment expectations, increase active participation in decision making, reduce uncertainty about the appropriate course of action, and help patients reach decisions that are more aligned with their stated values.

ELIGIBILITY:
Inclusion Criteria:

Providers

* Providers must be a licensed professional, either a physician (MD) or a nurse practitioner (APN) in the Division of Developmental and Behavioral Pediatrics at Cincinnati Children's Hospital.
* Provider must regularly treat patients within the age range and for the diagnoses of interest in this study (Autism Spectrum Disorders).

Parents

* Participants must be a parent or legal guardian who self-identifies as the primary caregiver of a child or adolescent with Autism Spectrum Disorder cared for by an enrolled provider in the Division of Developmental and Behavioral Pediatrics at Cincinnati Children's Hospital.
* Participants must be able to speak and read English in order to complete the surveys

Children

* Child or adolescent must have a clinical diagnosis of Autism Spectrum Disorder including one of the following diagnoses: a) Pervasive Developmental Disorder (PDD), b) Asperger's Syndrome, c) Autism Spectrum Disorder, d) Autism, e) Infantile Autism
* Child or adolescent must be between the ages of 4 years 0 months and 15 years 11 months
* Child or adolescent must be scheduled for a follow up visit with a Developmental-Behavioral Pediatric provider enrolled in the study.

Exclusion Criteria:

-Parents who are unable to speak and read English are not eligible for the study.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict | At the end of the Day 1 (initial study) visit
  The primary outcome of interest for this study is decisional conflict as measured immediately at the end of the Day 1 initial study clinic visit. This measure will also be collected before the Day 1 visit to be able to compare pre- and post- visit levels of decisional conflict. Additionally, this measure will be collected 3 months after the Day 1 visit to determine levels of ongoing decisional conflict that parents of children with autism experience.
  This will be measured using the Decisional Conflict Scale. This is a validated 16-item questionnaire which reports on the uncertainty experienced when feeling uninformed about the alternatives, benefits and risks, unclear about personal values, or unsupported in making a choice.

SECONDARY OUTCOMES:
Parent-physician interaction | During the Day 1 (initial study) visit
  The OPTION scale (validated 12-item measure) will be used to score parent-physician interactions developing a treatment plan based on coding of audio or video recordings of the clinic visit.

OTHER OUTCOMES:
Parental Knowledge of Medications for Challenging Behaviors in ASD | At the end of the Day 1 (initial study) visit
  Assess parents' knowledge of medications for challenging ASD behaviors with an 18-item checklist developed for this study. This includes questions on general knowledge about the role of medication in ASD treatment and assesses caregiver expectations of whether medication might improve specific challenging behaviors.
Parenting Stress | Before or at the time of the Day 1 (initial study) visit and at the 3 month interval follow up
  Will be measured using the Parenting Stress Index- Short Form. This is a validated 36-item questionnaire pertaining to the demands of taking care of a child. It includes 3 subscales and a total score: parental distress, parent-child dysfunctional interaction, and difficult child.
Shared Decision Making | At the end of the Day 1 (initial study) visit
  Parental perception of shared decision making during the clinical encounter will be assessed using the CollaboRATE. This is a brief, 3-question survey that assesses parent-reported shared decision making.
Child Behavioral Symptoms | Before or at the time of the Day 1 (initial study) visit and 3 month interval follow up
  Child behavioral symptoms will be measured at the time of the Day 1 (initial study) visit and 3 months later using:
  1. The Child Behavior Checklist (CBCL) will be used to assess behavioral functioning by domains of treatment. The CBCL is a commonly used clinical and research measure. The 120 scale items map onto Diagnostic and Statistical Manual(DSM)-oriented scales and will be used as a standardized measure of behavioral symptoms.
  2. Aberrant Behavior Checklist (ABC): 58-item caregiver report form developed to assess maladaptive behaviors in individuals with developmental disabilities and commonly used to assess behavior in studies of children with ASD.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Anixt, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Frazier TW, Shattuck PT, Narendorf SC, Cooper BP, Wagner M, Spitznagel EL. Prevalence and correlates of psychotropic medication use in adolescents with an autism spectrum disorder with and without caregiver-reported attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2011 Dec;21(6):571-9. doi: 10.1089/cap.2011.0057. Epub 2011 Dec 13. PMID 22166171
- [Background] Nickels K, Katusic SK, Colligan RC, Weaver AL, Voigt RG, Barbaresi WJ. Stimulant medication treatment of target behaviors in children with autism: a population-based study. J Dev Behav Pediatr. 2008 Apr;29(2):75-81. doi: 10.1097/dbp.0b013e31815f24f7. PMID 18478626
- [Background] Blum NJ, Feldman HM, Barbaresi WJ, Schonfeld DJ, Hansen RL, Forrest CB. Research priorities for developmental-behavioral pediatrics: a DBPNet consensus study. J Dev Behav Pediatr. 2012 Jul;33(6):509-16. doi: 10.1097/DBP.0b013e31825a7101. PMID 22710856
- [Background] O'Connor AM, Llewellyn-Thomas HA, Flood AB. Modifying unwarranted variations in health care: shared decision making using patient decision aids. Health Aff (Millwood). 2004;Suppl Variation:VAR63-72. doi: 10.1377/hlthaff.var.63. PMID 15471770
- [Background] Fiks AG, Mayne S, Localio AR, Feudtner C, Alessandrini EA, Guevara JP. Shared decision making and behavioral impairment: a national study among children with special health care needs. BMC Pediatr. 2012 Sep 21;12:153. doi: 10.1186/1471-2431-12-153. PMID 22998626
- [Background] Stacey D, Bennett CL, Barry MJ, Col NF, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Legare F, Thomson R. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD001431. doi: 10.1002/14651858.CD001431.pub3. PMID 21975733
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] Fowler FJ Jr, Levin CA, Sepucha KR. Informing and involving patients to improve the quality of medical decisions. Health Aff (Millwood). 2011 Apr;30(4):699-706. doi: 10.1377/hlthaff.2011.0003. PMID 21471491
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Brinkman WB, Hartl J, Rawe LM, Sucharew H, Britto MT, Epstein JN. Physicians' shared decision-making behaviors in attention-deficit/hyperactivity disorder care. Arch Pediatr Adolesc Med. 2011 Nov;165(11):1013-9. doi: 10.1001/archpediatrics.2011.154. PMID 22065181
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Brinkley J, Nations L, Abramson RK, Hall A, Wright HH, Gabriels R, Gilbert JR, Pericak-Vance MA, Cuccaro ML. Factor analysis of the aberrant behavior checklist in individuals with autism spectrum disorders. J Autism Dev Disord. 2007 Nov;37(10):1949-59. doi: 10.1007/s10803-006-0327-3. Epub 2006 Dec 21. PMID 17186368
- [Background] Zaidman-Zait A, Mirenda P, Zumbo BD, Georgiades S, Szatmari P, Bryson S, Fombonne E, Roberts W, Smith I, Vaillancourt T, Volden J, Waddell C, Zwaigenbaum L, Duku E, Thompson A; Pathways in ASD Study Team. Factor analysis of the Parenting Stress Index-Short Form with parents of young children with autism spectrum disorders. Autism Res. 2011 Oct;4(5):336-46. doi: 10.1002/aur.213. Epub 2011 Aug 31. PMID 21882359
- See also: Shared Decision Aid — http://www.autismspeaks.org/science/resources-programs/autism-treatment-network/tools-you-can-use/medication-guide